CLINICAL TRIAL: NCT06101355
Title: Comparison of the Effectiveness of Telerehabilitation in Individuals With Total Knee Arthroplasty
Brief Title: Effectiveness of Telerehabilitation in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Sema Nur Aslan, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Telerehabilitation
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Telerehabilitation; Home Exercise; Osteoarthritis; Orthopaedic Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group Based on Home Exercises (Experimental): Intervention group is home exercise program supplemented with visual and video resources using telerehabilitation.
  Interventions: Other: Telerehabilitation
- Standard Home Exercise Group (Active Comparator): Standard home based exercise group
  Interventions: Other: Standard Home Based Exercise Group

INTERVENTIONS:
Other: Telerehabilitation — Intervention group is home exercise program supplemented with visual and video resources using telerehabilitation. With the exercises, there will be video links, exercise visuals, and written explanations. Videos and visuals of the exercises recorded by the physiotherapist and uploaded to the Rehab My Patient application.
  Digital exercise forms will be prepared through the Rehab My Patient application. The intervention group will receive exercises, which prepared from the Rehab My Patient application ,digitally through WhatsApp. In this group, exercise sessions will be conducted with the physiotherapist once a week through video calls. Additionally, there will be one instance of messaging and one phone call for follow-up. Video calls and messaging will be conducted through WhatsApp.
  Arms: Telerehabilitation Group Based on Home Exercises
Other: Standard Home Based Exercise Group — Control group, standard home exercise program group , will receive the program as brochures. Although there will be no video supplement, the brochure will include visuals of the exercises. The control group will be monitored through three weekly voice calls.
  Arms: Standard Home Exercise Group

SUMMARY:
In patients who have had joint replacement surgery, there is a shortage of concrete evidence regarding the effectiveness of telerehabilitation. The aim of this study is to compare telerehabilitation with home based exercise program and standard home exercise program in total knee arthroplasty.

DETAILED DESCRIPTION:
The primary aim of our study is to assess the effectiveness of telerehabilitation in comparison to the conventional approach, specifically focusing on particular parameters, in the context of post-total knee arthroplasty surgery. This investigation will entail a comparative analysis between a home exercise program prescription supplemented with visual and video resources using telerehabilitation and the conventional home exercise program prescription.

The aim of our study is comparison between two exercise prescription modalities : a standard home exercise program and an internet-based program utilizing the Rehab My Patient software with visual and video support, in addition to telerehabilitation program, which involves exercise prescription oversight via video consultations. This comparison will include the following parameters : range of motion, proprioception , function, kinesiophobia, pain , patient adherence, patient satisfaction and Quadriceps muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 50 and over
* Having a primary total knee arthroplasty surgery
* To possess a device, such as a smartphone or tablet, that enables access to mobile applications.
* To have the capability to use the internet and to have internet access.
* Proficiency in reading and writing in the Turkish language
* Having a Mini-Mental State Examination(MMSE) score of 24 or higher
* To be willing to participate in the study

Exclusion Criteria:

* Having cognitive problem
* Having a secondary total knee arthroplasty surgery
* Havig a revision surgery
* Having a history of cerebrovascular and/or cardiovascular events in the last 3 months
* Having uncontrolled diabetes and/or hypertension
* Having a arthrogenic muscle inhibition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Flexion Range of Motion of the Knee | Postoperatively first day, fourth week and eight week
  Assessment of active and passive flexion range of motion of both knee with digital goniometer

SECONDARY OUTCOMES:
Demographic Data | Postoperatively first day
  The demographic data such as gender,age, body weight and height, comorbidities of the individuals included the study will be recorded
Mental State | Postoperatively first day
  Mini Mental State Examination consists of 30 questions.The test results range from 0 to 30 points. A score of 0-10 points indicates severe impairment, 10-20 points suggests moderate impairment, 20-25 points indicate mild impairment, and a score of 25-30 points is considered normal.
Range of Motion | Postoperatively first day, fourth week and eight week
  Assessment of range of motion of the knee including active and passive flexion and extension by digital goniometer
Assessment of Pain | Postoperatively first day, fourth week and eight week
  Assessment the pain while rest, night and activity by using Visual Analog Scale which is a 100 mm line drawn laterally on an A4 sheet of paper. The left end of the line shows "no pain at all", the right end shows "my pain is as bad as it could be", while the remaining part shows the intermediate values.
Assessment of Kinesiophobia | Postoperatively first day, fourth week and eight week
  Assessment of kinesiophobia via Brief Fear of Movement. This scale consists of 6 items, which are items 1, 2, 9, 10, 14, and 15 from the Tampa Scale for kinesiophobia. It is a valid approach for assessing movement fear in patients with osteoarthritis
Assessment of Artificial Joint Awareness | Postoperatively fourth week and eight week
  Assessment of artificial joint awareness via Forgotten Joint Score-12. This scale consists of 12 items.Item 12 of the scale has not been considered suitable for use in the Turkish population. High scores reflect the degree to which one can forget and adapt to the side of the surgery, typically represented as a percentage
Assessment of Pain, Stiffness and Physical Function | Postoperatively first day, fourth week and eight week
  Assessment of pain, stiffness and physical function via WOMAC(The Western Ontario and McMaster Universities). The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores indicates higher disability.
Assessment of Patient Adherence | Postoperatively fourth week and eight week
  Assessment of patient adherence via The Exercise Adherence Rating Scale. The scale consists of three sections: Part A, Part B, and Part C. Part A and Part B each consist of 6 questions, while Part C comprises 10 items.The total score ranges from 0 to 64. A high score indicates better adherence to exercise or a higher level of exercise compliance.
Assessment of Function | Postoperatively first day, fourth week and eight week
  5 Times Sit to Stand Test
Assessment of Telemedicine Satisfaction and Usefulness | Postoperatively fourth week and eight week
  Assessment of Telemedicine Satisfaction and Usefulness via Telemedicine Satisfaction and Usefulness Questionnaire(TSUQ). TSUQ consists of 21 items.This questionnaire assesses the satisfaction levels and usability of telemedicine services among individuals. The total score range from 21 to 105.
Assessment of Quadriceps Muscle Strength | Postoperatively fourth week and eight week
  Assessment of Quadriceps Muscle Strength via Lafayette Manual Muscle Tester.The Lafayette Manual Muscle Tester is used for the objective evaluation of muscle strength. It has both intra-rater and inter-rater reliability and is an ideal tool for tracking progress throughout the rehabilitation process.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Nur Aslan, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)